CLINICAL TRIAL: NCT05217823
Title: Long-term Stability of Er:YAG Laser Non-surgical Periodontal Treatment
Brief Title: Er:YAG Laser Treatment of Moderate Chronic Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Plovdiv Medical University (Other)
Responsible Party: Principal Investigator, Blagovesta Yaneva, Principle Investigator, Plovdiv Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Er:YAG - chronic periodontitis
Record Dates: First submitted 2022-01-04; First posted 2022-02-01 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Chronic Periodontitis, Generalized, Moderate
Keywords: Lasers; Periodontitis; Root planing; Treatment outcome
MeSH Terms: conditions — Chronic Periodontitis; Lymphoma, Follicular; Periodontitis | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Er:YAG laser (Experimental): Teeth treated with Er:YAG laser
  Interventions: Device: Er:YAG laser
- Hand instruments (Active Comparator): Teeth treated with Gracey curettes
  Interventions: Other: hand instruments

INTERVENTIONS:
Device: Er:YAG laser
  Other Names: Er:YAG laser, LiteTouch, Light Instruments, Israel
  Arms: Er:YAG laser
Other: hand instruments
  Other Names: Gracey curettes
  Arms: Hand instruments

SUMMARY:
The Er:YAG laser possesses specific characteristics allowing to be used in non-surgical periodontal treatment. The aim of the resent study was to evaluate the long-term clinical effectiveness of Er:YAG laser monotherapy in the treatment of moderate chronic periodontitis and to compare it with conventional hand instrumentation.

MATERIALS AND METHODS: 451 teeth (1,099 periodontal pockets) from 30 patients with moderate chronic periodontitis (initial probing pocket depth 4 to 6 mm) were allocated for subgingival scaling and root planing in two groups - hand instrumentation (control) and Er:YAG laser instrumentation with 100mJ/15Hz (test). Using a computerized periodontal probe, patients were examined for probing pocket depth (PPD), gingival recession (GR), clinical attachment level (CAL), bleeding on probing (BOP), plaque presence (FMPS) at baseline, one, three, six and 12 months after instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* at least two teeth per quadrant with PPD between 3,6 mm and 6,4 mm;
* loss of clinical attachment up to 4 mm
* bleeding on probing

Exclusion Criteria:

* periodontal treatment in the last 12 months;
* systemic diseases;
* systemic medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Probing pocket depth | 1 year
  Change in PPD (measured as a distance between the gingival margin and the depth of the pocket) using computerised periodontal probe

SECONDARY OUTCOMES:
Gingival recession | 1 year
  Change in GR (measured as a distance between the gingival margin and the cement-enamel junction) using computerised periodontal probe
Clinical attachment level | 1 year
  Change of CAL (measured as a distance between the cement-enamel junction and the depth of the pocket) using computerised periodontal probe
Bleeding on probing | 1 year
  Change in BoP
Plaque level | 1 year
  Change of Plaque index

IPD SHARING:
Plan to Share IPD: Undecided